CLINICAL TRIAL: NCT05934825
Title: A Multicenter Phase I/II Clinical Trial, Randomized, Double Blind, Controlled With Placebo to Evaluate Safety and Efficiency of Allogenic Adult Mesenchymal Stem Cells From Adipose Tissue in the Treatment of Draining Fistulas in Patients With Hidradenitis Suppurativa
Brief Title: Clinical Trial to Evaluate Safety and Efficiency of Mesenchymal Stem Cell in Patients With Hidradenitis Suppurativa
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Andalusian Network for Design and Translation of Advanced Therapies (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HidraQureS/2020
Record Dates: First submitted 2023-03-17; First posted 2023-07-07 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-07

CONDITIONS: Hidradenitis Suppurativa
MeSH Terms: conditions — Hidradenitis Suppurativa

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Injectable suspension of allogeneic adult mesenchymal stem cells (Experimental): Patients will receive an injectable suspension of allogeneic adult mesenchymal stem cells from adipose tissue intralesionally.
  Interventions: Biological: Injectable suspension of allogeneic adult mesenchymal stem cells
- Placebo (Placebo Comparator): Patients will receive the cell-free suspension vehicle: 49% DMEM without phenol red, 1% L-Alanine LGlutamine and 50% hyaluronic acid
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Injectable suspension of allogeneic adult mesenchymal stem cells — Cell therapy treatment will be administered in a single dose at the beginning of the study. The treatment consists of the administration of a single dose of allogeneic adult mesenchymal stem cells from adipose tissue. The dose is 120 million cells (drug volume: 20 ml, concentrated at 6 million cels/ml).
  Arms: Injectable suspension of allogeneic adult mesenchymal stem cells
Other: Placebo — The placebo consists of the administration of the excipient of the suspension without cells. The excipient is a mixture of 50% hyaluronic acid, 49% DMEM without phenol red and 1% L-Alanine-L Glutamine.
  Arms: Placebo

SUMMARY:
Multicenter Phase I/II Clinical Trial to Evaluate Safety and Efficiency of Allogenic Adult Mesenchymal Stem Cell from Adipose Tissue in Patients With Hidradenitis Suppurativa

ELIGIBILITY:
Inclusion Criteria:

* Patients who give informed consent for participation in the clinical trial
* Diagnosed 6 months before inclusion
* Drainage fistula with a minimum of 1 subcutaneous tract and 1 cutaneous drainage orifice evaluated clinically and by cutaneous ultrasound. The fistula must have active drainage 4 weeks prior to inclusion
* Treatment with Adalimumab for at least 12 weeks.
* Normal renal function or moderate chronic renal insufficiency with creatinine clearance values greater than 60 ml/min or serum creatinine less than 1.5 times the upper limit.
* Normal liver function with total bilirubin values less than 1.5 times the upper limit of normal and transaminases < 2.5 times the upper limit of normal.
* Hemogram and coagulation studies within normal values (Leukocytes ≥ 3000, Neutrophils ≥ 1500, Platelets ≥ 100000, hemoglobin>10g/dl).
* Negative blood pregnancy test for patients of childbearing age
* Acceptance by the patient, of childbearing age, to use safe contraceptive methods throughout the study, including six months of follow-up.
* Willingness and ability to comply with the visit schedule, treatment plan, clinical tests and all study procedures. and all study procedures.

Exclusion Criteria:

* Poorly controlled HS requiring additional systemic treatment or change of baseline anti-inflammatory therapy
* Abscess or inflammatory collection > 2 cm adjacent to the fistula to be treated.
* Previous surgical treatment on the draining fistula
* Known history of alcohol abuse in the 6 months prior to study entry
* Active malignancy or patients with a history of a previous malignant tumor.
* Presence or recent history of severe, progressive and uncontrolled hepatic, hematologic, gastrointestinal, endocrine, pulmonary, cardiac, neurologic, psychiatric or skin disease
* Congenital or acquired immunodeficiencies
* Positive serology for HIV, HCV or HBV.
* Active COVID-19 infection confirmed by serology and PCR or rapid antigen test
* Allergy to any of the components/excipients of the Investigational Product
* Major surgery or severe trauma in the previous 6 months
* Patients unwilling or unable to comply with study procedures.
* Anticipated need for surgery in the anatomical area for a reason other than hidradenitis suppurative
* Contraindication to the anesthetic procedure
* Systemic immunomodulatory biologic therapy other than Adalimumab, topical or systemic antibiotics for HS, systemic or intralesional corticosteroids, live vaccines, or any experimental treatment or intervention study participation.
* Contraindication of nuclear magnetic resonance with contrast.
* Women who are pregnant, breastfeeding, or of childbearing age who are not using an effective contraceptive method.
* Patients who are currently participating or have completed participation in a clinical trial in a period of less than 3 months or who have participated in an Advanced Therapies clinical trial at any previous time and have been assigned to an experimental group.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-10-26 (Actual); Primary Completion 2025-10-26 (Estimated); Study Completion 2025-10-26 (Estimated)

PRIMARY OUTCOMES:
Safety of the administration of allogeneic mesenchymal stem cells derived from adipose tissue assessed by Adverse Event Rate | 24 months
  To determine the safety of intralesional administration of allogeneic mesenchymal cells in draining fistulas in patients with hidradenitis suppurativa
Efficacy of the administration of allogeneic mesenchymal stem cells derived from adipose tissue assessed by Survival Rate | 23 months
  To evaluate the efficacy of intralesional administration of human allogeneic mesenchymal cells versus the control group, in terms of combined remission of the draining fistula.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Virgen de Las Nieves, Granada, Spain